CLINICAL TRIAL: NCT05795868
Title: The Effect of Compression Stockings on the Complaints, Well-Being and Sleep Quality of Pregnant Women With Restless Legs Syndrome
Brief Title: The Effect of Compression Stockings on the Complaints of Pregnant Women With Restless Leg Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Ozlem Kaplan, Reserch Asistant, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 221S452
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Restless Legs Syndrome; Pregnancy Related; Sleep Disorder
MeSH Terms: conditions — Restless Legs Syndrome; Sleep Wake Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Compression stockings group (Experimental): Pregnant women in the compression stockings group will wear the socks given for 3 weeks.
  Interventions: Device: Compression stocks
- Placebo sock group (Placebo Comparator): Pregnant women in the placebo socks group will wear the socks given for 3 weeks.
  Interventions: Other: Knee socks

INTERVENTIONS:
Device: Compression stocks — Pregnant women in the compression stockings group will wear the socks given for 3 weeks.
  Arms: Compression stockings group
Other: Knee socks — Pregnant women in the Knee socks group will wear the socks given for 3 weeks.
  Arms: Placebo sock group

SUMMARY:
The aim of this project is to determine the effect of compression stockings on the complaints, well-being and sleep quality of pregnant women with restless legs syndrome (RLS). The research is a pretest-posttest randomized placebo-controlled experimental study. The study will be carried out with a total of 70 people, 35 in the compression stocking group and 35 in the placebo stocking group. Study data will be collected with RLS Diagnostic Criteria Questionnaire Form, Research Criteria Compliance Form, Personal Information Form, RLS Severity Rating Scale, Pittsburgh Sleep Quality Index (PUKI), WHO-5 and Implementation Satisfaction Form. Pregnant women in both groups will wear the stockings given for three weeks after the first interview.

Data analysis obtained in the research will be performed in TURCOSA statistical software (Turcosa Analytics Ltd Co, Turkey, www.turcosa.com.tr).In comparisons, a value of p <0.05 will be considered statistically significant. In order to conduct the study, the necessary Academic Committee decision, Ethics Committee approval (December 08, 2021 and number 2021/781) and institutional permission were obtained. The individuals included in the study will be informed about the purpose of the research, their verbal consent will be obtained and the participant's informed consent form will be signed.

ELIGIBILITY:
Inclusion Criteria:

1. Least literate,
2. Between the ages of 18 and 40,
3. At 27 and above gestational week,
4. Single pregnancy,
5. Presence of RLS according to the RLS Diagnostic Criteria Questionnaire Form,
6. Having a severity of 11 and above according to the RLS Severity Rating Scale,
7. Using Iron, Vitamin D, Magnesium and Calcium,
8. Pregnant women with a hemoglobin level of 11 g/dl and above,
9. Pregnant women who can wear socks all day long, except for going to sleep, will be included in the study.

Exclusion Criteria:

1. Having a communication barrier,
2. Having a risky pregnancy (risk of preterm labor, cervical insufficiency, preeclampsia, polyhydramnios, macrosomic baby, etc.),
3. Having RLS before pregnancy,
4. Having a chronic disease (Diabetes, hypertension, thyroid, cardiovascular disease, etc.),
5. With maternal obesity (BMI>30)
6. Having sleep apnea before pregnancy,
7. Having any psychiatric disease and using antipsychotic and antidepressant drugs,
8. Using heparin, antihistamine, antiemetic, calcium channel blocker, dextromethorphan and decongestant type drugs,
9. Having a dermatological problem in the feet and legs,
10. Pregnant women with varicose veins on their feet and legs will not be included in the study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Since the study will be conducted with pregnant women with restless legs syndrome, only women were included in the study.
Enrollment: 70 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
RLS Severity Rating Scale | Change from baseline score at the end of 21. days
  The RLS Severity Rating Scale was developed in 2003 by the International Restless Legs Syndrome Study Group. The scale was applied in the selection of patients and in the weekly evaluation of RLS severity. The scale comprised ten questions; each question was scored between 0 and 4. Questions 1, 2, 4, 6, 7, and 8 were related to RLS symptoms, questions 5, 9, and 10 were related to the effect of the disease on the mental state and daily social activities of patients with RLS, and question 3 was about the diagnostic criteria of RLS. The overall score indicated the RLS severity. A minimum score of 0 and a maximum score of 40 could be obtained. A score between 1 and 10 corresponded to "mild," 11-20 "moderate," 21-30 "severe," and 31-40 "very severe" RLS.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | Change from baseline score at the end of 21. days
  The form consists of a total of 24 questions. Each question is scored between 0 and 3. Pittsburgh Sleep Quality Index score in the 0-21 range, with high scores indicating poor sleep quality. If the Pittsburgh Sleep Quality Index global score is greater than 5, it indicates that the sleep quality is significantly worse. The fact that the Pittsburgh Sleep Quality Index score is above 5 indicates that the person has serious trouble in at least two areas related to his sleep, or that he has mild or moderate difficulty in more than three areas.

OTHER OUTCOMES:
World Health Organization-5 Index of Well-being (WHO-5) | Change from baseline score at the end of 21. days
  The WHO-5 questionnaire consists of 5 items containing positive statements about the participant's feelings in the last 2 weeks. Each item is evaluated on a 6-point Likert-type scale between 0-5; 0 points indicates no positive feelings in the last 2 weeks, 5 points indicates continuous positive feelings. The raw score is calculated by adding the numbers from the five answers. The total score that can be obtained from the scale varies between 0 and 25. 0 represents the worst possible quality of life and 25 the best possible quality of life, while a score below 13 indicates poor quality of life.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Özlem Kaplan, Kayseri
  - Erciyes University, Kayseri

IPD SHARING:
Plan to Share IPD: No
Will be shared after the study ends.

REFERENCES:
- [Derived] Kaplan O, Baser M, Ozgun MT. The effect of compression stockings on the complaints well-being and sleep quality of pregnant women with restless legs syndrome: a randomized controlled study. Rev Assoc Med Bras (1992). 2024 Aug 16;70(7):e20240145. doi: 10.1590/1806-9282.20240145. eCollection 2024. PMID 39166663